CLINICAL TRIAL: NCT03715530
Title: A Comparison of the Measurement of Placental Alpha-microglobulin-1 in Cervicovaginal Discharge, Sterile Speculum Exam, and Amniodye Testing for the Diagnosis of Preterm Premature Rupture of Membranes
Brief Title: Use of Placental Alpha Microglobulin-1(PAMG-1) to Diagnose Premature Rupture of Membranes in Pregnant Women
Acronym: PAMG-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection has halted due to no further assays provided by AmniSURE
Sponsor: Mark Santillan (Other)
Collaborators: AmniSure International LLC (Other)
Responsible Party: Sponsor-Investigator, Mark Santillan, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 200706757
Record Dates: First submitted 2018-10-16; First posted 2018-10-23 (Actual); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Preterm Labor; Preterm Birth
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Pregnant subjects (Experimental): These are pregnant women that are admitted to Labor &Delivery (L&D) or an outpatient in the Women's Health Clinic that are being evaluated for rupture of membranes.
  Interventions: Device: PAMG-1 immunoassay
- Pregnant controls (Active Comparator): These women will be found primarily in the Women's Health Clinic, when being seen for their routine antepartum appointments. Most of them will be recruited at about 36 weeks, since they will be having a pelvic exam at this time, as part of their routine antepartum care.
  Interventions: Device: PAMG-1 immunoassay
- Non pregnant controls (Sham Comparator): These women will be found in the Women's Health Clinic, when being seen for gynecology appointments. Nursing staff and the dashboard will help to identify those patients who will be having a pelvic exam.
  Interventions: Device: PAMG-1 immunoassay

INTERVENTIONS:
Device: PAMG-1 immunoassay — The procedure includes the insertion of a PAMG-1 swab into the subject's vaginal vault without a speculum for one minute. Once the swab is obtained, the treating physician will place the swab in a solvent vial for one minute. A developing strip is then placed in a vial and allowed to develop for five minutes. The results are read from the developing strip.

SUMMARY:
The study is to evaluate the accuracy of a test device called "PAMG-1" to see if a pregnant women has ruptured membranes in comparison to standardly used testing methods.

DETAILED DESCRIPTION:
The study is to evaluate the accuracy of the PAMG-1 immunoassay in comparison to standard diagnostic methods for premature preterm rupture of membranes including the sterile speculum exam and the amniodye test as the gold standard.

The procedure includes the insertion of a swab into the subject's vaginal vault without a speculum for one minute. Once the swab is obtained, the treating physician will place the swab in a solvent vial for one minute. A developing strip is then placed in a vial and allowed to develop for five minutes. The results are read from the developing strip. Processing of this swab will be performed without further involvement of the study participant. The insertion of the swab is a one time procedure and is the only addition to any standard of care that would applied to the patient during their clinical evaluation at that time. Given the study group and both pregnant and non-pregnant controls, standard of care procedures will include a wide variety of obstetrical and/or gynecological (OB/Gyn) procedures including but not limited to a vaginal exams, sterile speculum exams (including pap smears), biopsies, and amniocentesis. The swab for the PAMG-1 immunoassay will be performed after other evaluations are performed. Medical records of the subject and (if applicable) her newborn infant will be reviewed for data pertaining to the study, including, but not limited to, maternal and fetal outcomes at the time of enrollment and after delivery and history of the present illness requiring an OB/Gyn evaluation. The study participants will not be asked to do anything in addition to what is expected for the swab and their clinical visit. The PAMG-1 immunoassay will be obtained during the subjects regularly scheduled clinic appointment or hospital visit. No follow appointments will be needed.

ELIGIBILITY:
Inclusion Criteria:

* women 18 to 50 years of age
* being seen at the University of Iowa Women's Healthcare Clinic

Exclusion Criteria:

* men

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Santillan, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnant Subjects | Pregnant Controls | Non Pregnant Controls
Started | 33 | 42 | 87
Completed | 30 | 41 | 85
Not Completed | 3 | 1 | 2
Not completed — Lost to Follow-up | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnant Subjects | Pregnant Controls | Non Pregnant Controls | Total
Number analyzed (Participants) | 33 | 42 | 87 | 162
Age, Continuous [Mean (Full Range); unit: years] | 25.7 [18 to 37] | 29.2 [19 to 42] | 31.2 [18 to 49] | 29.6 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 42 | 87 | 162
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 31 | 41 | 86 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 5 | 9
  White | 30 | 34 | 79 | 143
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PAMG-1 Test Results That Matched the Results of Gold Standard Testing
Description: Number of participants with PAMG-1 test results that matched the results of gold standard testing
Time Frame: The assessment of the accurance PAMG-1 is completed by the end of the first study visit; one day.
Measure: Number; unit: participants
Arm/Group | Pregnant Subjects | Pregnant Controls | Non Pregnant Controls
Number analyzed (Participants) | 30 | 41 | 85
participants | 27 | 41 | 83

ADVERSE EVENTS:
Arm/Group | Pregnant Subjects | Pregnant Controls | Non Pregnant Controls
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/42 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/42 | 0/87
Other Adverse Events (participants affected / at risk) | 0/33 | 0/42 | 0/87

LIMITATIONS AND CAVEATS:
Data collection has halted due to no further assays provided by AmniSURE.

No statistical analysis was completed at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes